CLINICAL TRIAL: NCT00597181
Title: A Clinical Study Comparing the Inflammatory Response of the Ex-Press Mini Glaucoma Shunt to Trabeculectomy in Subjects With Open-Angle Glaucoma
Brief Title: A Clinical Study Comparing the Inflammatory Response of the Ex-Press Mini Shunt to Trabeculectomy
Acronym: Optonol
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Patient population limited
Sponsor: Indiana University (Other)
Collaborators: Optonol (Unknown)
Responsible Party: Louis B. Cantor, M.D., Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0710-28
Record Dates: First submitted 2008-01-07; First posted 2008-01-17 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Glaucoma
Keywords: Inflammatory response
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Trabeculectomy with Mitomycin C 0.2 mg/cc for 2 minutes
  Interventions: Procedure: Trabeculectomy with mitomycin c
- 2 (Active Comparator): Ex-Press mini shunt; Model R50 with mitomycin C 0.2 mg/cc for 2 minutes
  Interventions: Procedure: Ex-Press mini shunt with mitomycin c

INTERVENTIONS:
Procedure: Trabeculectomy with mitomycin c — mitomycin c 0.2 mg/cc for 2 minutes
  Arms: 1
Procedure: Ex-Press mini shunt with mitomycin c — mitomycin c 0.2 mg/cc for 2 minutes
  Arms: 2

SUMMARY:
The less invasive nature of the Ex-Press Mini shunt with mitomycin C induces less post-operative inflammation than trabeculectomy with mitomycin c.

DETAILED DESCRIPTION:
The purpose of this study is to quantify the degree of post-operative inflammation in eyes which have undergone either trabeculectomy filtering surgery or Ex-Press mini shunt insertion. Early intraocular pressure control and postoperative complications will also be noted.

ELIGIBILITY:
Inclusion Criteria:

All subjects must:

1. Be willing and able to provide written Informed Consent.
2. Be able and willing to follow instructions on the use of post- operative medication and likely to complete the entire course of the study.
3. Be male or female of any race at least 18 years of age.
4. Have medically uncontrolled glaucoma for which they have elected to undergo surgery.
5. Diagnosed with primary open angle glaucoma, pigmentary or pseudoexfoliation glaucoma.

Exclusion Criteria:

No subject may:

1. Have any contraindication to intraocular surgery.
2. Diagnosed with: primary angle closure glaucoma, normal tension glaucoma, secondary glaucoma, neovascular glaucoma.
3. Have any active ocular disease other than glaucoma that would interfere with study parameters (such as: uveitis, ocular infection, or severe dry eye). Subjects with mild chronic blepharitis, age-related macular degeneration and background diabetic retinopathy may be enrolled at the discretion of the investigator.
4. Have laser ALT or SLT within the past 3 months or cataract surgery within the last six months.
5. Require use of ocular NSAID or systemic steroids.
6. Have known allergy or sensitivity to mitomycin C
7. Have corneal abnormalities that would interfere with the ability to obtain an adequate laser flare measurement.
8. Be concurrently enrolled in an investigational drug or device study or participation within the last 30 days in any investigational drug or device study.
9. Be pregnant, nursing, planning a pregnancy, or be of childbearing potential and not using a reliable form of contraception (a woman is considered of childbearing potential unless she is postmenopausal, has had a uterus and/or both ovaries removed, or has had a bilateral tubal ligation).
10. Have a situation or condition that in the investigator's opinion may put the subject at significant risk, may confound the study results, or may interfere significantly with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Aqueous humor flare | 2 months

SECONDARY OUTCOMES:
Aqueous humor cell | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Louis B Cantor, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- IU Eye at Carmel, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Hille K, Hans J, Manderscheid T, Spang S, Ruprecht KW. [Laser flare in combined cataract and glaucoma surgery]. Ophthalmologe. 2001 Jan;98(1):47-53. doi: 10.1007/s003470170199. German. PMID 11220271
- [Background] Maris PJ Jr, Ishida K, Netland PA. Comparison of trabeculectomy with Ex-PRESS miniature glaucoma device implanted under scleral flap. J Glaucoma. 2007 Jan;16(1):14-9. doi: 10.1097/01.ijg.0000243479.90403.cd. PMID 17224744
- [Background] Shah SM, Spalton DJ, Allen RJ, Smith SE. A comparison of the laser flare cell meter and fluorophotometry in assessment of the blood-aqueous barrier. Invest Ophthalmol Vis Sci. 1993 Oct;34(11):3124-30. PMID 8407220
- [Background] Dahan E, Carmichael TR. Implantation of a miniature glaucoma device under a scleral flap. J Glaucoma. 2005 Apr;14(2):98-102. doi: 10.1097/01.ijg.0000151688.34904.b7. PMID 15741808
- [Background] Shields, MB Textbook of Glaucoma. Fourth Edition; Williams & Wilkins, Baltimore, 1998.
- [Background] Guyer DR, Yannuzzi LA, Chang S, Shields JA, Green WR Retina-Vitreous-Macula. W.B. Saunders Company, Philadelphia, 1999.